CLINICAL TRIAL: NCT01941238
Title: Incidence of Hypoglycemia During Ramadan in Patients With Type1 Diabetes on Insulin Pump Versus Multi-dose Insulin Injection
Brief Title: Incidence of Hypoglycemia During Ramadan in Patients With Type1 Diabetes on Insulin Pump Versus Multi Dose Injection
Status: Completed | Type: Observational
Sponsor: Reem Mohammad Alamoudi (Other)
Responsible Party: Sponsor-Investigator, Reem Mohammad Alamoudi, Consultant Endocrinology, King Abdullah International Medical Research Center
Organization: King Abdullah International Medical Research Center (Other)
Other Study IDs: RE12-002
Record Dates: First submitted 2013-09-04; First posted 2013-09-13 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Type 1 Diabetes
Keywords: Ramadan; Fasting; Diabetes; Type1; Insulin; Pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Fasting; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Insulin pump
- MDI

SUMMARY:
Managing patients with type1 diabetes when fasting Ramadan is very challenging. Insulin pump offers the advantage of flexibility and precision to administering insulin and has been proven to reduce severe hypoglycemia compared to multi-dose injection (MDI). However, there are extremely limited studies on the difference between insulin pump compared to MDI on the incidence of hypoglycemia and other acute complications during fasting Ramadan

The investigators hypothesized that insulin pump would be associated with less hypoglycemic events during fasting Ramadan compared to MDI without deterioration in glycemic control. Results of this study are descriptive but will fill a current gap in knowledge and may contribute to development of future guidelines for the management of type1DM during Ramadan.

ELIGIBILITY:
Inclusion Criteria:

1. DM type 1
2. Age ≥14 years
3. Patients on insulin pump (more than 3 months)
4. Patients on MDI (glargine or detemir combined with aspart or lispro) regimen
5. Diagnosis of type 1 DM of more than 6 months.
6. Willing to do Self Monitoring Blood Sugar (SMBG)
7. Have no other contraindication to fast

Exclusion Criteria:

1. Patient with renal or hepatic impairment
2. Patient with diagnosed adrenal insufficiency
3. Pregnancy
4. Alcoholism
5. Any diagnosed psychiatric disease
6. Can not do SMBG

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population of our study is all patients with type1DM treated at three National Guard institutiuons in three different cities of Saudi Arabia (Riyadh, Alahsa, Dammam) with either insulin pump or MDI
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Incidence of hypoglycemia | 5 weeks
  Rates of hypoglycemia during fasting ramadan in insulin pump users and MDI users [Hypoglycemia defined as blood glucose level ≤ 70 mg/dl ( 3.9 mmol/l)]

SECONDARY OUTCOMES:
Number of fasting days lost | 5 weeks
  To estimate the number of days they needed to brake their fast due to acute complications (hypoglycemia, severe hyperglycemia, or DKA).
Glycemic control | Two (2) months
  To assess the glycemic control in the two groups using HbA1c and Fructosamine assays.
overnight hypoglycemia | 5 weeks
  To estimate the rates of overnight hyperglycemia in both groups.
Rate of acute complications | 5 weeks
  To estimate presence of severe hyperglycemia and /or DKA episodes in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- National Guards Hospital, Dammam, Saudi Arabia

REFERENCES:
- [Derived] Alamoudi R, Alsubaiee M, Alqarni A, Aljaser S, Saleh Y, Salam A, Eledrisi M. Attitudes and habits of patients with type 1 diabetes during fasting Ramadan. J Clin Transl Endocrinol. 2018 Sep 6;14:1-4. doi: 10.1016/j.jcte.2018.09.001. eCollection 2018 Dec. PMID 30294552